CLINICAL TRIAL: NCT06659237
Title: Fecal and Oral Microbiota Between Pancreatic Cancer and Benign/Low-grade Malignant Tumor Patients
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-PCAMICROBE-2
Record Dates: First submitted 2024-10-21; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-05

CONDITIONS: Microbiome; Pancreatic Neoplasms; 16s RRNA
Keywords: fecal microbiome; oral microbiome; pancreatic neoplasms; 16s rRNA
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 16S rRNA or shot-gun metagenomics of oral and fecal samples from patients with pancreatic neoplasms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pancreatic cancer: Patients pathologically diagnosed with cancer or high-grade mucinous tumors based on surgical specimens or puncture samples
  Interventions: Diagnostic Test: 16s rRNA or shotgun metagenomics
- Benign or low-grade malignant pancreatic tumor: Patients with pathological diagnoses such as low-grade intraductal papillary mucinous neoplasm (IPMN), mucinous cystadenoma, serous cystadenoma, chronic pancreatitis, neuroendocrine tumors, or solid pseudopapillary tumors
  Interventions: Diagnostic Test: 16s rRNA or shotgun metagenomics

INTERVENTIONS:
Diagnostic Test: 16s rRNA or shotgun metagenomics — 16s rRNA or shotgun metagenomics on oral and fecal samples

SUMMARY:
Significant gaps exist in understanding the gastrointestinal microbiota in patients with pancreatic cancer (PCA) versus benign or low-grade malignant pancreatic tumors (NPCA). This study aimed to analyze these microbiota characteristics and explore their potential use in distinguishing malignant pancreatic lesions.

DETAILED DESCRIPTION:
In the past decade, microbiome research has rapidly progressed, revealing the critical roles of fecal and oral microbiota in maintaining internal homeostasis. Studies employing 16S rRNA and metagenomics have highlighted dysbiosis of the fecal and oral microbiota as closely linked to PCA development and progression. However, significant gaps exist in understanding the fecal and oral microbiota in patients with pancreatic cancer (PCA) versus benign or low-grade malignant pancreatic tumors (NPCA). This study aimed to analyze fecal and oral microbiota characteristics, and to establish classifiers to discriminate PCA from NPCA, providing a reference for early clinical identification of malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pancreatic tumor detected via imaging with no prior treatment before sample collection
* Patients volunteer to provide oral and fecal samples

Exclusion Criteria:

* Current or previous diagnoses of (a) other malignancies, (b) infectious diseases, (c) oral or gastrointestinal disorders (d) psychiatric or neurodegenerative disorders
* Specific medical procedures or interventions within defined periods, including (a) antibiotic, hormone therapy, or immunosuppressant within the past three months, (b) gastrointestinal reconstructive surgery within the past three months, (c) frequent use of cathartics, antidiarrheals, or therapeutic doses of probiotics within the past month, (d) oral or gastrointestinal examinations within the past three days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a pancreatic tumor detected via imaging
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
the accuracy of the diagnostic classifier | From enrollment to the end of treatment at 8 weeks
  we used random forest algorithm to construct oral and fecal microbiome classifiers to discriminate PCA and NPCA. AUC value was used to evaluate the efficacy of the classifiers

CONTACTS AND LOCATIONS:
Overall Officials: Menghua Dai, MD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Department of General Surgery, Peking Union Medical College Hospital (PUMCH), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No